CLINICAL TRIAL: NCT05751187
Title: Pembrolizumab Plus Bevacizumab and Chemotherapy as First-Line Treatment for Advanced or Metastatic Non-Squamous NSCLC Patients With EGFR Exon 20 Insertion Mutation: An Open-Label, Single-Arm, Phase II Trial
Brief Title: Pembrolizumab Plus Bevacizumab and Chemotherapy for Non-Squamous NSCLC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Baohui Han, Professor, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS22087
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Non-squamous NSCLC
Keywords: EGFR exon 20 insertion
MeSH Terms: interventions — pembrolizumab; Bevacizumab; Pemetrexed; Cisplatin; Carboplatin; Folic Acid; Vitamin B 12; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Bevacizumab + Chemotherapy (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin Area Under the Curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4-6 cycles followed by pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression.
  Interventions: Biological: Pembrolizumab; Biological: Bevacizumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Dietary Supplement: Folic acid 350-1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4 mg

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab was given as 200 milligrams (mg) via intravenous (IV) infusion over 30 minutes on Day 1 of each 21-day cycle.
Biological: Bevacizumab — Bevacizumab was given as 15 mg/kg via intravenous (IV) infusion on Day 1 of each 21-day cycle.
Drug: Pemetrexed — Pemetrexed was given as 500 mg/m^2 via intravenous (IV) infusion (with vitamin supplementation) on Day 1 of each 21-day cycle for 4-6 cycles.
Drug: Cisplatin — Cisplatin was given as 75 mg/m^2 via intravenous (IV) infusion (administered approximately 30 minutes after pemetrexed infusion) on Day 1 of each 21-day cycle for 4-6 cycles.
Drug: Carboplatin — Carboplatin was given as Aare Under the Curve (AUC) 5 (5 mg/mL/min; over 15-60 min) via intravenous (IV) infusion (administered immediately after pemetrexed infusion) on Day 1 of each 21-day cycle for 4-6 cycles.
Dietary Supplement: Folic acid 350-1000 μg — Orally; at least 5 doses of folic acid must be taken during the 7 days preceding the first dose of pemetrexed, and folic acid dosing must continue during the full course of therapy and for 21 days after the last dose of pemetrexed.
Dietary Supplement: Vitamin B12 1000 μg — Intramuscular injection in the week preceding the first dose of pemetrexed and once every 3 cycles thereafter. Subsequent vitamin B12 injections may be given on the same day as pemetrexed administration.
Drug: Dexamethasone 4 mg — For prophylaxis; orally twice per day (or equivalent). Taken the day before, the day of, and the day after pemetrexed administration.

SUMMARY:
This study is designed to evaluate the efficacy and safety of Pembrolizumab in combination with Bevacizumab and chemotherapy in advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) with EGFR exon 20 insertion mutation.

ELIGIBILITY:
Inclusion Criteria:

1. According to the 8th edition of the AJCC/UICC TNM staging system for NSCLC, patients with locally advanced (stage III B/III C), metastatic or recurrent (stage IV) nonsquamous NSCLC confirmed by histology or cytology who are unable to undergo surgery and radical concomitant radiochemotherapy and are confirmed to have at least one measurable lesion according to RECIST 1.1.
2. Patients harboring exon 20 insertions detected by ARMS or NGS or other approved methods.
3. Age ≥18 years and ≤75 years.
4. ECOG PS score: 0 to 1
5. Have a life expectancy of at least 3 months.
6. Have not received prior systemic treatment including chemotherapy, checkpoint inhibitors, TKIs, and anti-angiogenesis agents for their advanced/metastatic NSCLC. Subjects who received adjuvant or neoadjuvant therapy including immunotherapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of advanced/metastatic disease. Palliative radiotherapy must be completed 7 days before the first dose of study drugs and participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
7. Have adequate organ function as defined in the following： (1) Adequate bone marrow function Absolute neutrophil count(ANC) ≥ 1500/uL; Platelets≥10x104/uL; Hemoglobin ≥9.0g/dL or ≥5.6 mmol/L; (2) Adequate kidney function Creatinine≤ 1.5 x upper normal limit (ULN), OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥30 mL/min for the participant with creatinine levels >1.5 × institutional ULN (3) Adequate liver function Total bilirubin ≤ 1.5 x upper normal limit (ULN) OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN; Aspartate Aminotransferase (AST) (SGOT) ≤ 2.5 xULN (≤ 5.0 x ULN if hepatic metastases); Alanine Aminotransferase (ALT) (SGPT) ≤ 2.5 x ULN (≤ 5.0x ULN if hepatic metastases); (4) Coagulation function International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless the participant is receiving anticoagulant therapy as long as PT or aPTT is within the therapeutic range of intended use of anticoagulants.
8. A male participant must agree to use contraception during the treatment period and plus an additional 90 days (a spermatogenesis cycle) for study treatments after the last dose of study treatment and refrain from donating sperm during this period; A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and plus 30 days (a menstruation cycle) for study treatments after the last dose of study treatment.
9. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
10. Archival tumor tissue sample or newly obtained [core, incisional, or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin-embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
11. For hepatitis B-positive subjects:

(1) Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have an undetectable HBV viral load prior to enrollment.

(2) Participants should remain on anti-viral therapy throughout the study intervention and follow local guidelines for HBV anti-viral therapy post-completion of the study intervention.

(3) Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening.

(4) Participants must have completed curative anti-viral therapy at least 4 weeks prior to enrollment.

Exclusion Criteria:

1. Small cell lung cancer (including mixed small cell and non-small cell lung cancer);
2. Patients who have received systemic treatment for advanced/metastatic disease especially have received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g, CTLA-4, OX 40, CD137);
3. Patients concurrently with 19del or 21L858R or other mutation types located in exon 18-21
4. Patients who are known to have active brain metastases diagnosed by CT or MRI at the time of screening, however, participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without the requirement of steroid treatment for at least 14 days prior to the first dose of the study intervention.;
5. Patients with severe and/or uncontrolled diseases, such as:

(1) Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmias; uncontrolled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); (2) Active or uncontrolled serious infection; (3) Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; (4) Not completely controlled eye inflammation or eye infection, or any condition that may lead to the above-mentioned ocular diseases (5) Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L); (6) Routine urine test result indicates that urine protein ≥++, and 24-hour urine protein quantitation is confirmed to be > 1.0 g; (7) Active tuberculosis, etc.; (8) Uncontrolled hypercalcemia (> 1.5 mmol/L calcium ion or calcium > 12 mg/dL or corrected serum calcium > ULN), or symptomatic hypercalcemia requiring continued diphosphate therapy; (9) Long-term unhealed wounds or fractures; 6. Patients who have a history of psychotropic drug abuse and cannot abstain from it or have mental disorders; 7. Patients who are known to have severe allergies (≥ grade 3) to active ingredients and any excipients of pembrolizumab 8. Patients who have other malignant tumors (except radical cervical carcinoma in situ, non-melanoma skin cancer, etc.) at the same time; patients who are evaluated by the investigator to have concomitant diseases that seriously endanger the safety of the patients or affect the patients completing the study.

9. The subjects or their sexual partners cannot or refuse to take effective contraceptive measures during the clinical trial 10. Pregnant or breast-feeding women 11. Patients in other situations who are evaluated by the investigator to be ineligible to be enrolled; 12. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of the study intervention. Administration of killed vaccines is allowed (such as COVID-19 vaccines).

13. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study drug.

14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.

15. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.

16. Has a known history of Human Immunodeficiency Virus (HIV) infection. 17. Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.

18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

19. Has had an allogeneic tissue/solid organ transplant. 20. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to administration of pembrolizumab.

21. Patients who have contraindications of antiangiogenic therapy, including the presence of cavities, and bleeding tendencies judged by the treating physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 24 months
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per Response Criteria in Solid Tumors version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 24 months
  PFS is defined as the time from the first dose of study treatment to the first documented progressive disease (PD) per Response Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on blinded independent central review (BICR), or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of ≥1 new lesion was also considered PD.
Overall Survival (OS) | Up to approximately 24 months
  OS was defined as the time from the first dose of study treatment to death due to any cause.
Duration of Response (DOR) | From time of first documented evidence of CR or PR to Up to approximately 24 months
  For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from the first documented evidence of a CR or PR until PD or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. DOR assessments were based on BICR with confirmation. The DOR per RECIST 1.1 for all participants who experienced a confirmed CR or PR is presented.
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 24 months
  An AE was defined as any untoward medical occurrence in a participant-administered study treatment that did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE is presented.
Number of Participants Who Discontinued Any Study Drug Due to an AE | Up to approximately 24 months
  The number of participants who discontinued any randomized study drug due to an AE is presented.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

REFERENCES:
- [Background] Chen K, Pan G, Cheng G, Zhang F, Xu Y, Huang Z, Fan Y. Immune microenvironment features and efficacy of PD-1/PD-L1 blockade in non-small cell lung cancer patients with EGFR or HER2 exon 20 insertions. Thorac Cancer. 2021 Jan;12(2):218-226. doi: 10.1111/1759-7714.13748. Epub 2020 Nov 18. PMID 33210451
- [Background] Dong ZY, Zhang JT, Liu SY, Su J, Zhang C, Xie Z, Zhou Q, Tu HY, Xu CR, Yan LX, Li YF, Zhong WZ, Wu YL. EGFR mutation correlates with uninflamed phenotype and weak immunogenicity, causing impaired response to PD-1 blockade in non-small cell lung cancer. Oncoimmunology. 2017 Jul 26;6(11):e1356145. doi: 10.1080/2162402X.2017.1356145. eCollection 2017. PMID 29147605
- [Background] Lu S, Wu L, Jian H, Chen Y, Wang Q, Fang J, Wang Z, Hu Y, Sun M, Han L, Miao L, Ding C, Cui J, Li B, Pan Y, Li X, Ye F, Liu A, Wang K, Cang S, Zhou H, Sun X, Ferry D, Lin Y, Wang S, Zhang W, Zhang C. Sintilimab plus bevacizumab biosimilar IBI305 and chemotherapy for patients with EGFR-mutated non-squamous non-small-cell lung cancer who progressed on EGFR tyrosine-kinase inhibitor therapy (ORIENT-31): first interim results from a randomised, double-blind, multicentre, phase 3 trial. Lancet Oncol. 2022 Sep;23(9):1167-1179. doi: 10.1016/S1470-2045(22)00382-5. Epub 2022 Jul 28. PMID 35908558